CLINICAL TRIAL: NCT07246603
Title: Virtual Housecalls: Redesigning Pediatric Primary Care Adolescent Obesity Treatment
Acronym: VHC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM300000084; R01DK144911 (NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Class I Obesity; Pediatric Obesity
Keywords: Lifestyle Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors and MPIs will be masked to treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Housecalls Intervention (VHC) (Experimental): Includes standard in-person pediatric primary care, 6 months of telehealth sessions with a behavior coach (3 months with weekly sessions, 3 months with bi-weekly sessions), and weekly exercise videos sent electronically for the 6 month intervention. Sessions include real-time skill building that uses items or space in families' home to tailor the treatment and personalize content application to their context.
  Interventions: Behavioral: Virtual Housecalls
- Enhanced Treatment as Usual (TAU+) (No Intervention): Includes standard in-person pediatric primary care, enhanced with PPCP training on obesity treatment guidelines and publicly available education regarding healthy eating and exercise, delivered to participants on a contact schedule matched to the intervention group.

INTERVENTIONS:
Behavioral: Virtual Housecalls — 26 contact hours of evidence-based intensive health and behavioral lifestyle treatment, as per the American Academy of Pediatrics Clinical Practice Guidelines
  Arms: Virtual Housecalls Intervention (VHC)

SUMMARY:
This pragmatic randomized clinical trial tests a novel intensive health behavior and lifestyle intervention, conducted via telehealth, to treat class I adolescent obesity in pediatric primary care. Results will inform scalable approaches that meet the recommended treatment dose and effectively treat obesity in this setting.

DETAILED DESCRIPTION:
This trial will test Virtual Housecalls (VHC) in a pragmatic randomized clinical trial with 250 adolescents ages 12-15 years with class 1 (non-severe) obesity (BMI≥95% and <120% of the 95%) and a participating parent/caregiver (N=250 dyads / 500 individuals). VHC includes 26 hours of treatment, by combining in-person PPCP visits (every 3m) with 6m of virtual visits conducted by a behavior coach (3m weekly, 3m every 2 weeks), and weekly exercise videos. The control arm will receive enhanced treatment as usual (TAU+), which includes usual care by their pediatric primary care practitioner (PPCP), augmented with publicly available education, sent on an attention-matched contact schedule. All PPCPs will receive training on the AAP Clinical Practice Guideline for obesity treatment and reports of participant progress at 3, 6, and 12m. Assessments of anthropometrics, dietary intake, physical activity, parenting and the home environment will be completed at 0, 3, 6 (post-intervention), and 12m (maintenance), with the primary endpoint at 6m. The investigators will evaluate the efficacy of VHC on adolescent change in body mass index (primary outcome) and dietary and physical activity behaviors (secondary outcomes). Investigators will also evaluate how treatment dose impacts BMI reduction.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* English or Spanish-speaking
* 12-15 years of age
* Receiving care at a participating clinic
* Body Mass Index (BMI) ≥95% and <120% of the 95%
* Access to a mobile device with a webcam that can receive texts

Parent Inclusion Criteria:

* English or Spanish-speaking
* Primary legal guardian ≥18 years of age living with the adolescent

Exclusion Criteria:

* conflicts that would inhibit the ability to participate in all aspects of the study as outlined in the study protocol
* family plans to move outside of the study area or plans to no longer be a patient at a participating clinic in the 12 month study period
* the primary care provider or PI determines that the study is not clinically or medically appropriate (e.g., significant psychiatric, cognitive, physical or developmental conditions that would impair their ability to complete assessments, participate in study sessions, or conduct physical activity) based on screening at study onset
* adolescent exhibits severe dietary restriction or compensatory behavior (e.g., vomiting, laxative abuse) based on screening at study onset and clinical interview by a study psychologist
* adolescent is currently pregnant/plans to become pregnant during study period
* adolescent is participating in another weight loss program, has had or plans to undergo weight loss surgery
* adolescent has a chronic medical condition(s) and/or uses medication that substantially impacts or interferes with growth, appetite, weight or physical activity participation
* adolescents taking anti-obesity medication are ineligible if they are not a stable dose for at least 3 months prior to study participation

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) Change | 0 - 6 months
  Adolescent height (cm) and weight (kg) will be measured in triplicate by trained staff wo are masked to treatment assignment. Height and weight values will be used to calculate Body Mass Index (BMI) specific to age and sex using the Centers for Disease and Control reference data.

SECONDARY OUTCOMES:
Body Mass Index (BMI) Maintenance | 6 - 12 months
  Adolescent height (cm) and weight (kg) will be measured in triplicate by trained staff wo are masked to treatment assignment. Height and weight values will be used to calculate Body Mass Index (BMI) specific to age and sex using the Centers for Disease and Control reference data.
Energy Intake | 0-6-months, 6-12-months
  Dietary intake (kilocalories/day); total of 1, 24-hour recall per assessment time point. Recalls will be obtained using the Automated Self-Administered 24-hour (ASA-24) dietary assessment tool with the assistance of trained staff who are masked to treatment assignment. Assessment time points include baseline (0), 6-month, and 12-months.
Diet Quality | 0-6-months, 6-12-months
  The Healthy Eating Index (HEI) will be used to measure diet quality using 1, 24-hour recall per assessment time point. Recalls will be obtained using the Automated Self-Administered 24-hour (ASA-24) dietary assessment tool with the assistance of trained staff who are masked to treatment assignment. HEI scores will be calculated from the ASA-24 recall data. Assessment time points include baseline (0), 6-month, and 12-months.
Physical Activity | 0-6-months, 6-12-months
  The Physical Activity Questionnaire for Adolescents (PAQ-A) will assess changes in time spent participating in moderate to vigorous physical activity (MVPA).
Treatment Dose | 0-6-months
  Treatment dose(s) (number and contact time) to yield Body Mass Index (BMI) reductions will be explored. Treatment dose includes all intervention components: 1) parent-teen dyad sessions, 2) parent-only sessions, 3) exercise videos, and 4) standard of care medical visits with pediatric provider.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Bean, PhD, Principal Investigator — Virginia Commonwealth University; Shari Barkin, PhD, Principal Investigator — Emory University
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States

IPD SHARING:
Plan to Share IPD: No